CLINICAL TRIAL: NCT02953977
Title: Strong Men, Strong Communities: Cultural Tradition to Improve Native Men's Health
Brief Title: Strong Men, Strong Communities Diabetes Risk Reduction in American Indian Men
Acronym: SMSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Denise Dillard, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DK102728-01A1 (NIH)
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Block randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Intervention (Experimental): Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program
- Delayed Intervention (Other): Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — An adapted version of the Diabetes Prevention Program will be delivered to intervention participants.

SUMMARY:
SMSC will inform the design and implementation of culturally informed, community-based lifestyle interventions for diabetes prevention in AI men in our partner communities and elsewhere, as well as in men of other minority groups who experience a heavy burden of diabetes.

DETAILED DESCRIPTION:
American Indian (AI) males experience profound health disparities compared to their counterparts in all other U.S. racial and ethnic groups. AI men have the highest age-adjusted prevalence of type 2 diabetes (~18%) among U.S. men, while non-Hispanic White men have the lowest (~7%). In recent decades, AIs have seen a disproportionate increase in diabetes-related complications and mortality compared to all other groups, such that age-adjusted diabetes death rates in AI men are now almost twice those in White men.

Several large randomized, con trolled trials in non-AIs confirm that type 2 diabetes can be prevented or delayed by interventions that promote healthy lifestyles, but little empirical data exist on interventions to prevent diabetes in AI men. In the clinic-based U.S. Diabetes Prevention Program (DPP), only 55 out of 3,234 participants were AI men. Similarly, in the diabetes prevention programs in Native communities, participation by AI males is low, ranging from 33% to 74%. Many explanations have been posited for the low participation rates among men of all races in lifestyle interventions. Recruiting AI men in clinic-based programs is difficult because they tend to seek clinical care less often than women. AI men's perceptions of normative health behaviors and gender roles may also discourage participation, particularly in mixed-gender groups. Therefore, an urgent need exists for diabetes risk reduction programs tailored to the unique values and habits of AI men, with a particular focus on recruitment and retention

ELIGIBILITY:
Inclusion Criteria:

* Must be male and self-reported American Indian; ages 18-75, A BMI ≥25 kg/m2 and/or a waist circumference >90 cm for men; no prior diabetes diagnosis; No history of heart disease, serious illness, cancer diagnosis in the last five years, or other conditions that may impede or prohibit participation; reliable internet access; access to a computer, tablet, or smartphone; have an active email address; and, willingness to consent to randomization

Exclusion Criteria:

* Females, under 18 years old or older than 75 years

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males or individuals who identify as male
Enrollment: 257 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline weight | 6 months
  7.5% weight loss from baseline weight

SECONDARY OUTCOMES:
Change in dietary habits and consumption and frequency of physical activity | 6 months
  Dietary change using the NCI Fat & Veg Screener and Fruit Screener
Changes in Stages of Change for healthy eating and physical activity | 12 months
  Transtheoretical model of stage of change for weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- IREACH, Seattle, Washington, United States

REFERENCES:
- [Result] Sinclair K, Gonzales K, Woosley C, Cree TR, Garza CM, Buchwald D. An Intersectional Mixed Methods Approach to Understand American Indian Men's Health. Int J Mens Soc Community Health. 2020;3(2):e66-e89. doi: 10.22374/ijmsch.v3i2.35. Epub 2020 Sep 8. PMID 34485829
- [Result] Sinclair K, Carty C, Gonzales K, Nikolaus C, Gillespie L, Buchwald D. Strong Men, Strong Communities: Design of a Randomized Controlled Trial of a Diabetes Prevention Intervention for American Indian and Alaska Native Men. Am J Mens Health. 2020 Jul-Aug;14(4):1557988320945457. doi: 10.1177/1557988320945457. PMID 32757825